CLINICAL TRIAL: NCT05638295
Title: A Randomized Phase II Study of AMG 510 (Sotorasib) With or Without Panitumumab in Advanced Solid Tumors: A ComboMATCH Treatment Trial
Brief Title: Testing the Use of AMG 510 (Sotorasib) and Panitumumab as a Targeted Treatment for KRAS G12C Mutant Solid Tumor Cancers (A ComboMATCH Treatment Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-09876; NCI-2022-09876 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY191-E5 (Other: ECOG-ACRIN Cancer Research Group); EAY191-E5 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2022-12-02; First posted 2022-12-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Panitumumab; sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort I Arm A (sotorasib, panitumumab) (Experimental): Patients receive sotorasib PO QD on days 1-28 and panitumumab IV on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples, biopsy, and CT or MRI on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Panitumumab; Drug: Sotorasib
- Cohort I Arm B (sotorasib) (Active Comparator): Patients receive sotorasib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may cross-over to cohort II. Patients also undergo collection of blood samples, biopsy, and CT or MRI on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Sotorasib
- Cohort II (sotorasib, panitumumab) (Experimental): Patients receive combination therapy as in Arm A.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Panitumumab; Drug: Sotorasib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; E7.6.3; Human IgG2K Monoclonal Antibody; MoAb ABX-EGF; MoAb E7.6.3; Monoclonal Antibody ABX-EGF; Monoclonal Antibody E7.6.3; Vectibix
  Arms: Cohort I Arm A (sotorasib, panitumumab); Cohort II (sotorasib, panitumumab)
Drug: Sotorasib — Given PO
  Other Names: AMG 510; AMG-510; AMG510; Lumakras; Lumykras

SUMMARY:
This phase II ComboMATCH treatment trial tests how well AMG 510 (sotorasib) with or without panitumumab works in treating patients with KRAS G12C mutant solid tumors that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Sotorasib is in a class of medications called KRAS inhibitors. It works by blocking the action of the abnormal protein that signals cancer cells to multiply. This helps stop or slow the spread of cancer cells. Panitumumab is in a class of medications called monoclonal antibodies. It works by slowing or stopping the growth of cancer cells. Giving combination panitumumab and sotorasib may kill more tumor cells in patients with advanced solid tumors with KRAS G12C mutation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of the combination of AMG 510 (sotorasib) and panitumumab as compared to AMG 510 (sotorasib) alone in patients with advanced/metastatic KRAS G12C mutated solid tumors (except colorectal carcinoma [CRC] and non-small cell lung carcinoma [NSCLC]) as measured by progression free survival (Cohort 1).

II. To evaluate the efficacy of the combination of AMG 510 (sotorasib) and panitumumab in patients with advanced/metastatic KRAS G12C mutated solid tumors that have progressed on a prior KRAS G12C inhibitor as measured by response rate (Cohort 2).

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of the combination of AMG 510 (sotorasib) and panitumumab as compared to AMG 510 alone in patients with advanced/metastatic KRAS G12C mutated solid tumors (except CRC and NSCLC) as measured by response rate, disease control rate, and overall survival (Cohort 1).

II, To evaluate the efficacy of the combination of AMG 510 (sotorasib) and panitumumab in patients with advanced/metastatic KRAS G12C mutated solid tumors that have progressed on a prior KRAS G12C inhibitor as measured by disease control rate, progression free survival (PFS), and overall survival (Cohort 2).

III. To further evaluate the safety and tolerability of the combination of AMG 510 (sotorasib) and panitumumab.

IV. To collect tissue and provide it to the ComboMATCH Registration Protocol to assess concordance between the diagnostic tumor mutation profile generated by the Designated Laboratories, the pre-treatment biopsy mutation profile, and the pre-treatment circulating tumor-derived deoxyribonucleic acid (DNA) (ctDNA) mutation profile from plasma, as described in ComboMATCH Registration Protocol.

CORRELATIVE EXPLORATORY OBJECTIVES:

I. To investigate the impact of concomitant mutations on the clinical benefit. II. To evaluate if changes in circulating tumor DNA (ctDNA) over time correlate with response to treatment.

III. To evaluate the relative mutant allele fraction of KRAS mutation as a predictor of clinical benefit.

IV. To evaluate if ERK 1/2 and PI3K pathway activation correlate with response and/or resistance.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients who have never received a KRAS G12C inhibitor are randomized to arms A or B.

ARM A: Patients receive sotorasib orally (PO) once daily (QD) on days 1-28 and panitumumab intravenously (IV) on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples, biopsy, and computed tomography (CT) or magnetic resonance imaging (MRI) on study.

ARM B: Patients receive sotorasib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may cross-over to cohort II. Patients also undergo collection of blood samples, biopsy, and CT or MRI on study.

COHORT II: Patients who have received a KRAS G12C inhibitor are assigned to arm C.

ARM C: Patients receive combination therapy as in Arm A.

After completion of study treatment, patients are followed up at 30 days and then every 3-6 months for up to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto EAY191 and must have been given a treatment assignment to ComboMATCH to EAY191-E5 based on the presence of an actionable mutation as defined in EAY191
* Patient must be enrolled on the ComboMATCH Registration Protocol (EAY191) at the time of registration/randomization to the EAY191-E5 study
* Patient must be >= 18 years of age
* Patient must have a KRAS G12C alteration as determined by the ComboMATCH screening assessment
* Patient must have disease that can be safely biopsied and agree to a pre-treatment biopsy or have tissue available from within 12 months prior to the date of registration on the ComboMATCH Registration Trial (EAY191-E5)

  * NOTE: The current actionable marker of interest (aMOI)/actionable alteration list for this treatment trial can be found on the Cancer Trials Support Unit (CTSU) website: www.ctsu.org (final URL pending)
  * NOTE: Novel/Dynamic aMOI can be submitted for review per the process described in the ComboMATCH registration protocol
* Patient must have cytologically/histologically confirmed advanced/metastatic solid tumor
* Patient must have progressed on at least one line of standard of care therapy in the advanced/metastatic setting

  * NOTE: Patients who have progressed on a prior human epidermal growth factor receptor (EGFR) inhibitor will meet this criterion
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 (or Karnofsky performance status >= 60%)
* Patient must have at least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) documented by imaging obtained within 28 days prior to registration/randomization
* Patient must not have any serious active infection within 4 weeks prior to EAY191-E5 registration/randomization (e.g., requiring hospitalization and/or intravenous [IV] antibiotics) or currently receiving oral or IV antibiotics for the treatment of infection. Patients receiving prophylactic antibiotics are eligible
* Patient must have the ability to retain oral medication and not have any clinically significant gastrointestinal abnormalities that might alter absorption
* Patient must not have any history of or current evidence of non-infectious interstitial lung disease (ILD)/pneumonitis
* Patient must not have a history of allergic reactions attributed to either of the study agents or to agents of similar chemical or biologic composition
* Patient must have completed full treatment cycle 21 days prior to EAY191-E5 registration/randomization if they have received prior chemotherapy, biological cancer therapy, radiation therapy or an investigational agent/device. Patients must have recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade 1 or better from any adverse events due to prior cancer therapy (with the exception of alopecia)
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. All patients of childbearing potential must have a blood test or urine study within 14 days prior to registration/randomization to rule out pregnancy. A patient of childbearing potential is defined as anyone, regardless of whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and for at least 6 months after the last dose of protocol treatment. Patients must not breastfeed while receiving protocol treatment and for one week (7 days) after the last dose of AMG 510 (sotorasib) and 2 months after the last dose of panitumumab
* Patients must not have neuropathy ≥ grade 2 within 14 days prior to registration/randomization
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Human immunodeficiency virus (HIV)-infected patients no effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac history, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trail, patients should be class 2B or better
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (obtained ≤ 28 days prior to protocol registration/randomization)
* Aspartate aminotransferase (AST) (serum (glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase ([SGPT]) < 3 x institutional upper limit of normal (obtained ≤ 28 days prior to protocol registration/randomization)
* Creatinine =< 1.5 x institutional ULN OR creatinine clearance > 50 mL/min/1.73 m^2 for patients with creatinine levels > 1.5 mg/dL as per Cockcroft-Gault (obtained ≤ 28 days prior to protocol registration/randomization)
* COHORT I: Patient must not have colorectal cancer or non-small cell lung cancer
* COHORT I: Patient must not have been previously treated with a KRAS G12C inhibitor
* COHORT II: Patient must have progressed after treatment at the recommended phase II dose (RP2D) of any KRAS G12C inhibitor

  * NOTE: Patients on cohort 1 who experience progression on Regimen 2 (AMG 510 [sotorasib] alone) may be eligible to enroll on cohort 2 and receive combination treatment with panitumumab and AMG 510 (sotorasib). Patients must meet performance status requirements and laboratory values as above and must be begin treatment within 7 days of enrollment. Migration to cohort 2 must take place within 6 months of progression, with no intervening anti-cancer therapy given.
  * NOTE: Cohort migration following disease progression is dependent on a slot being available. MATCHBox makes the new treatment assignment following initiation of a step 2 registration for this treatment trial
* COHORT II: Patient must not have been previously treated with a KRAS G12C inhibitor in combination with an EGFR inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) (Cohort I) | From registration to documented disease progression or death from any cause, assessed up to 3 years
  PFS will be compared between the arms using a one-sided log rank test with 10% type I error. Cox's proportional hazards model will be used to estimate the PFS hazard ratio between the treatment arms and a two-sided 80% confidence interval will be reported (to correspond to the one-sided 10% type I error). Confidence intervals on most other quantities will use the two-sided 90% level.
Best objective response (Cohort II) | From the start of the treatment until disease progression/recurrence, assessed up to 3 years
  Will be evaluated using the criteria defined by Response Evaluation Criteria in Solid Tumors) version 1.1 for patients with solid tumors.
Overall response rate (ORR) (Cohort II) | From the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 3 years
  The exact 90% confidence interval on the ORR (determined using the method of Atkinson and Brown) will be reported. If the number of analyzable cases is less than 35, a 5% one-sided test will still be used.

SECONDARY OUTCOMES:
Overall survival (OS) (Cohort I) | Up to 3 years
  OS distributions by treatment will be estimated and 90% confidence intervals on estimated rates at 6 and 12 months will be reported. The OS hazard ratio will be estimated using Cox proportional hazards model and a 90% confidence interval reported.
ORR (Cohort I) | Up to 3 years
  Will be compared using Fisher's exact test and exact 90% confidence intervals for the rates in each arm will be computed.
Disease control rates (Cohort I) | From the start of the treatment until the criteria for progression are met, assessed up to 3 years
  Will be compared using Fisher's exact test and exact 90% confidence intervals for the rates in each arm will be computed.
PFS (Cohort II) | At 6 and 12 months, assessed up to 3 years
  Will be estimated and 90% confidence intervals on estimated rates will be reported.
OS (Cohort II) | At 6 and 12 months, assessed up to 3 years
  Will be estimated and 90% confidence intervals on estimated rates will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen R Spencer, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (181):
- United States (181):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Outpatient Center - Oak Lawn, Oak Lawn, Illinois
  - Advocate High Tech Medical Park, Palos Heights, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Regional Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Medical Center-First Hill, Seattle, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm